CLINICAL TRIAL: NCT05773898
Title: Contribution of Psychological Autopsy to the Understanding of Suicidal Behaviors in French Overseas Territories
Acronym: AUTOPSOM
Status: Recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Department for Research, Studies, Evaluation and Statistics, French Health and Social Affairs Ministry, France (Unknown); French National Institute for Health and Medical Research, MOODS Unit (Unknown); Clinical research and Innovation Office, Martinique (Unknown); SOS KRIZ, Martinique (Unknown); Amiens University Hospital, France (Unknown); Suicide Prevention Resource Center, French Guiana (Unknown); Cayenne Hospital Center, French Guiana (Unknown); University Hospital, La Réunion (Unknown); Tahiti Hospital Center, French Polynesia (Unknown); Regional Health Agency, Martinique (Unknown); Regional Health Agency, French Guiana (Unknown); Regional Health Agency, La Somme (Unknown); Regional Health Agency, La Réunion (Unknown)
Responsible Party: Sponsor
Other Study IDs: 22_RIPH3_14; 2022-A02413-40 (Other: French National Medicines and Health Products safety Agency)
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Suicide; Mental Disorders; Prognostic Factors
Keywords: Suicide; Psychological autopsies; epidemiology; risk factors; psycholinguistic approach; French overseas territories
MeSH Terms: conditions — Suicide; Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- person close to the deceased: Relatives will be invited to participate in two semi-structured research interviews in the form of a storytelling interview with an interviewer. All interviews will be conducted after obtaining the participants' non-objection. The interviews will be recorded and, once transcribed, will be analysed.
  Interventions: Other: other

INTERVENTIONS:
Other: other — The interviewers will collect data from relatives using questionnaires and evaluation grids based on an identification form, a Life Trajectory questionnaire, an anthropological evaluation grid, a retrospective psychiatric diagnosis questionnaire (SCID), a socio-demographic questionnaire, a questionnaire on suicide risks and a questionnaire on emotional state.

SUMMARY:
The mains objectives of our project are to coordinate the monitoring of suicides and to identify common or specific suicide risk factors in four overseas DROM-COM (French Polynesia, La Reunion, French Guiana and Martinique) by comparing to a site in mainland France (Amiens). A mixed approach (quantitative and qualitative) will be used, based on semi-directed interviews of the psychological autopsy type.

DETAILED DESCRIPTION:
Epidemiological studies on suicide are rare in Overseas France. Nevertheless, studies conducted independently in New Caledonia (NC) and French Guiana were able to highlight a high prevalence of suicides in minority indigenous populations (Kanaks and Amerindians). These data therefore suggest a socio-cultural variability of suicides within the different territories. Psychological autopsies (used in NC) are an innovative approach that has already proven worldwilde its effectiveness in researching socio-cultural factors and prevalence of mental disorders in suicide subjects (Inserm). However, the qualitative analysis of psychological autopsies, even if it is very complete, is limited to known factors of suicide risk. Given the ethnic specificities of suicidal behavior and the socio-cultural richness of each overseas territory, an exploratory anthropologic approach will make it possible to complete identification of risk factors for suicide or combinations of these specific factors (profiles).

Our project will improve the data collection of suicide cases with the implementation of a network in each site (Public Health Department, Emergency units, Coroner offices, GP, associations, families…). Then interview with proxies of subjects deceased by suicide will allow psychological autopsy (questionnaires SCID to detect mental disorders, Life Trajectories, to detect life events and their burden, Anthropologic for socio-cultural aspects and Psycholinguistic analysis).

The total duration of the project will be 24 months with the recruitment of a maximum of 30 cases per site. Duration of the inclusion period will be 23 months, duration of follow-up per participant 1 month. The follow-up interview will be carried out one month after the inclusion interview. It will make it possible to establish a post-vention of suicide among the bereaved and an evaluation of the impact of the psychological autopsy interviews and the life trajectories of the bereaved.

ELIGIBILITY:
Inclusion Criteria:

* Persons close of the deceased
* Persons who knew about his/her childhood
* Age 18 or over
* Interviewed for the study between 2 and 11 months after the suicide

Exclusion Criteria:

* People with neuropsychiatric disorders that may affect the quality of the information collected, cognitive (memory and expression) and judgmental functions
* People who refuses to participate
* Persons referred to articles L.1121-6, L.1121-7, L. 1121-8 L.1121-1-2 of the French Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to the relatives of a person who died by suicide.
  The deceased had been living for at least two years in one of the five study territories and information on cause of death information was obtained from potential sources on suicide victims.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Existence of risk factors and mental disorders evaluated by Structured Clinical Interview for Diagnostic (SCID) | 1 month
  Number and percentage of mental disorders presented by the deceased and identified on the basis of data collected during DSM 5 diagnostic interviews.

SECONDARY OUTCOMES:
Assessment and comparison of risk factors and mental disorders | 1 month
  The number of risk factors identified and the number of mental disorders detected will be compared between the overseas territories and the Somme department.
Existence or not of violence in childhood or during life among suicide cases | 1 month
  The variables related to childhood violence will be presented with the number of subjects "n" expressed as a percentage.
Score of adversity by the Life Trajectory Questionnaire | 6 month
  Once the interviews have been completed, the recordings will be transcribed semi-automatically via the HappyScribe® online platform. The resulting verbatim recordings will then be used as data for psycholinguistic and anthropological analyses.
  The qualitative data will then be transformed into quantitative data following the methodology developed by Brown and Harris, in which a panel of experts (researchers from our team and clinicians) assigns an overall rating for each five-year period, according to the severity of the burden of adversity carried by the person. This rating, from 1 to 6, makes it possible to determine the burden of adversity in the development of the individual (detailed description Séguin et al, 2007). It is the ratings of adversity that will form the curve of these trajectories.
Existence of language, social and anthropological elements associated with suicide risk factors | 6 month
  an audio-recording will record responses to semi-structured interview using anthropological approach. After transcription, the qualitative data gained from these questions will be analyzed using thematic analysis to understand the main themes (Representations of mental illness and suicidal commitment. Religious beliefs and cultural practices. Use of traditional methods to treat mental illness).
  A part of the transcription will also be analyzed using psycholinguistic approach. The words will be defined according to their frequency of occurrence and the most frequent grouped according to several "reference universes" associated with central notions (e.g. feeling, sensation, behavior, time, family, crisis, suicide, etc.). The visualization of the reference universes will summarize the frequency and proximity of key words and will make it possible to obtain a cognitive and mental representation of the speech.

CONTACTS AND LOCATIONS:
Overall Officials: STEPHANE AMADEO, Pr, Principal Investigator — University hospital, Martinique
Locations (1):
- Centre Hospitalier Universitaire de Martinique - Hôpital Pierre ZOBDA QUITMAN, Fort-de-France, France, Martinique

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Amiot M, Amadeo S, Merle S, Guidere M, Jehel L, Seguin M, Spodenkiewicz M. Identifying suicidal risk factors in the French Overseas Territories with multimethod psychological autopsy (AUTOPSOM): a mixed-methods study protocol. BMJ Open. 2024 Jul 16;14(7):e079405. doi: 10.1136/bmjopen-2023-079405. PMID 39013644